CLINICAL TRIAL: NCT01657344
Title: Improving the Quality of Pediatric Emergency Care Using an Electronic Medical Record Registry and Clinician Feedback
Brief Title: PECARN Emergency Care Registry
Status: Completed | Type: Observational
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency); Pediatric Emergency Care Applied Registry Network (PECARN) (Unknown)
Responsible Party: Sponsor
Other Study IDs: 12-009177; R01HS020270-01A1 (AHRQ)
Record Dates: First submitted 2012-08-02; First posted 2012-08-06 (Estimated); Results first posted 2019-10-21 (Actual); Last update posted 2019-10-21 (Actual); Status verified 2019-09

CONDITIONS: Pediatric Emergency Care

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ED Patients: All patients (age 0-18 regardless of race, ethnicity, or gender and of diagnosis or chronic health condition) who are registered in the ED.

SUMMARY:
The objectives of this study are to: develop an emergency care visit registry for pediatric patients for Quality Improvement purposes and to support future research; to use the emergency care visit registry to collect stakeholder-prioritized emergency care performance improvement measures for important pediatric medical and trauma conditions; and report emergency care performance improvement measures.

ELIGIBILITY:
Inclusion Criteria:

* All patients (0-18) who registered in the ED

Exclusion Criteria:

* Greater than 18 years of age for ED patients

Max Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Study subjects are all patients (0-18 regardless of race, ethnicity, or gender and of diagnosis or chronic health condition) who are registered to the ED.
Sampling Method: Non-Probability Sample
Enrollment: 2019461 (Actual)
Dates: Start 2012-01 (Actual); Primary Completion 2017-07-20 (Actual); Study Completion 2017-07-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth R Alpern, MD, Principal Investigator — Ann & Robert H Lurie Children's Hospital of Chicago
Locations (5):
- United States (5):
  - The Children's Hospital of Colorado, Aurora, Colorado
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Data Coordinating Center, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes
When the study is completed, the data coordinating center (DCC) will prepare a distributable database in compliance with Federal requirements.This database will be de-identified sufficiently that it will not be subject to Federal regulations nor the Health Insurance Portability and Accountability Act (HIPAA).

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All participating sites' IRBs have granted a waiver of informed consent and assent for this study. In addition, all participating sites' IRBs have a granted a waiver of written authorization for HIPAA. Patients will not be approached for recruitment.
Groups:
- CHOP Base Emergency Department (ED) Patients; Cincinnati Children's Hospital Medical Center (CCHMC) Base ED; CCHMC Satellite ED; Children's National Medical Center (CNMC) Base ED; CNMC Satellite ED; The Children's Hospital Colorado Base ED; The Children's Hospital Colorado Satellite ED: All patients (age 0-18 regardless of race, ethnicity, or gender and of diagnosis or chronic health condition) who are registered in the ED in the calendar year of 2011 through 2021.
Period: Overall Study
Arm/Group | CHOP Base Emergency Department (ED) Patients | Cincinnati Children's Hospital Medical Center (CCHMC) Base ED | CCHMC Satellite ED | Children's National Medical Center (CNMC) Base ED | CNMC Satellite ED | The Children's Hospital Colorado Base ED | The Children's Hospital Colorado Satellite ED
Started | 421622 | 409967 | 196300 | 376517 | 157802 | 316477 | 140776
Completed | 421622 | 409967 | 196300 | 376517 | 157802 | 316477 | 140776
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Patients Visits to the Emergency Department: There are no arms for this study. We are collecting all electronic patient data for all patients that present to the Emergency Department. Quality performance measures are constructed directly from the data in the registry.
Arm/Group | Patients Visits to the Emergency Department
Number analyzed (Participants) | 2019461
Age, Customized [Median (Inter-Quartile Range); unit: years] — Median Age Population: Number Analyzed corresponds to the number of ED visits at each ED.
  years
    CHOP Base ED: number analyzed (Participants) | 421622
    CHOP Base ED | 4.9 [1.7 to 10.8]
    CCHMC Base ED: number analyzed (Participants) | 409967
    CCHMC Base ED | 5.6 [1.8 to 12.5]
    CCHMC Satellite ED: number analyzed (Participants) | 196300
    CCHMC Satellite ED | 5.6 [2.0 to 11.4]
    CNMC Base ED: number analyzed (Participants) | 376517
    CNMC Base ED | 4.8 [1.7 to 10.7]
    CNMC Satellite ED: number analyzed (Participants) | 157802
    CNMC Satellite ED | 4.4 [1.8 to 9.5]
    The Children's Hospital Colorado Base ED: number analyzed (Participants) | 316477
    The Children's Hospital Colorado Base ED | 5.6 [1.9 to 11.7]
    The Children's Hospital Colorado Satellite ED: number analyzed (Participants) | 140776
    The Children's Hospital Colorado Satellite ED | 4.8 [1.9 to 9.7]
Sex/Gender, Customized [Count of Participants; unit: Participants] — Population: The number of participants analyzed is equal to the number of ED visits for the hospital ED named for the row, not the overall study.
  Participants
    CHOP Base ED: number analyzed (Participants) | 421622
    CHOP Base ED: Female | 199620
    CHOP Base ED: Male | 221993
    CHOP Base ED: Missing | 9
    CCHMC Base ED: number analyzed (Participants) | 409967
    CCHMC Base ED: Female | 200281
    CCHMC Base ED: Male | 209672
    CCHMC Base ED: Missing | 14
    CCHMC Satellite ED: number analyzed (Participants) | 196300
    CCHMC Satellite ED: Female | 94879
    CCHMC Satellite ED: Male | 101416
    CCHMC Satellite ED: Missing | 5
    CNMC Base ED: number analyzed (Participants) | 376517
    CNMC Base ED: Female | 177254
    CNMC Base ED: Male | 199263
    CNMC Base ED: Missing | 0
    CNMC Satellite ED: number analyzed (Participants) | 157802
    CNMC Satellite ED: Female | 76526
    CNMC Satellite ED: Male | 81276
    CNMC Satellite ED: Missing | 0
    The Children's Hospital Colorado Base ED: number analyzed (Participants) | 316477
    The Children's Hospital Colorado Base ED: Female | 151354
    The Children's Hospital Colorado Base ED: Male | 165119
    The Children's Hospital Colorado Base ED: Missing | 4
    The Children's Hospital Colorado Satellite ED: number analyzed (Participants) | 140776
    The Children's Hospital Colorado Satellite ED: Female | 66164
    The Children's Hospital Colorado Satellite ED: Male | 74610
    The Children's Hospital Colorado Satellite ED: Missing | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: The number analyzed in the rows corresponds to each hospital's emergency department, rather than the overall participants.
  Participants
    CHOP Base ED: number analyzed (Participants) | 421622
    CHOP Base ED: American Indian/Alaskan Native | 259
    CHOP Base ED: Asian/Pacific Islander | 13411
    CHOP Base ED: Black | 257886
    CHOP Base ED: Other | 46347
    CHOP Base ED: White | 102105
    CHOP Base ED: Unknown | 221
    CHOP Base ED: Missing | 1393
    CCHMC Base ED: number analyzed (Participants) | 409967
    CCHMC Base ED: American Indian/Alaskan Native | 255
    CCHMC Base ED: Asian/Pacific Islander | 2632
    CCHMC Base ED: Black | 174845
    CCHMC Base ED: Other | 43551
    CCHMC Base ED: White | 181269
    CCHMC Base ED: Unknown | 7191
    CCHMC Base ED: Missing | 224
    CCHMC Satellite ED: number analyzed (Participants) | 196300
    CCHMC Satellite ED: American Indian/Alaskan Native | 170
    CCHMC Satellite ED: Asian/Pacific Islander | 2597
    CCHMC Satellite ED: Black | 24745
    CCHMC Satellite ED: Other | 31795
    CCHMC Satellite ED: White | 132981
    CCHMC Satellite ED: Unknown | 3936
    CCHMC Satellite ED: Missing | 76
    CNMC Base ED: number analyzed (Participants) | 376517
    CNMC Base ED: American Indian/Alaskan Native | 414
    CNMC Base ED: Asian/Pacific Islander | 4142
    CNMC Base ED: Black | 225581
    CNMC Base ED: Other | 49335
    CNMC Base ED: White | 33775
    CNMC Base ED: Unknown | 59908
    CNMC Base ED: Missing | 3362
    CNMC Satellite ED: number analyzed (Participants) | 157802
    CNMC Satellite ED: American Indian/Alaskan Native | 37
    CNMC Satellite ED: Asian/Pacific Islander | 93
    CNMC Satellite ED: Black | 153787
    CNMC Satellite ED: Other | 1567
    CNMC Satellite ED: White | 579
    CNMC Satellite ED: Unknown | 1316
    CNMC Satellite ED: Missing | 423
    The Children's Hospital Colorado Base ED: number analyzed (Participants) | 316477
    The Children's Hospital Colorado Base ED: American Indian/Alaskan Native | 1334
    The Children's Hospital Colorado Base ED: Asian/Pacific Islander | 9473
    The Children's Hospital Colorado Base ED: Black | 52847
    The Children's Hospital Colorado Base ED: Other | 86204
    The Children's Hospital Colorado Base ED: White | 158877
    The Children's Hospital Colorado Base ED: Unknown | 7597
    The Children's Hospital Colorado Base ED: Missing | 145
    The Children's Hospital Colorado Satellite ED: number analyzed (Participants) | 140776
    The Children's Hospital Colorado Satellite ED: American Indian/Alaskan Native | 507
    The Children's Hospital Colorado Satellite ED: Asian/Pacific Islander | 2308
    The Children's Hospital Colorado Satellite ED: Black | 1056
    The Children's Hospital Colorado Satellite ED: Other | 33179
    The Children's Hospital Colorado Satellite ED: White | 90715
    The Children's Hospital Colorado Satellite ED: Unknown | 12996
    The Children's Hospital Colorado Satellite ED: Missing | 15

OUTCOME MEASURES:

1. Primary Outcome: The Number of Visits Obtained From Electronic Health Record Data From the Sites
Description: The number of visits obtained from electronic health record data from the sites
Time Frame: January 2012 - June 2016
Measure: Number; unit: number of visits
Groups:
- CHOP Base Emergency Department (ED); Cincinnati Children's Hospital Medical Center (CCHMC) Base ED; CCHMC Satellite ED; Children's National Medical Center (CNMC) Base ED; CNMC Satellite ED; The Children's Hospital Colorado Base ED; The Children's Hospital Colorado Satellite ED: All ED visits from patients (age 0-18 regardless of race, ethnicity, or gender and of diagnosis or chronic health condition) who are registered in the ED.
Arm/Group | CHOP Base Emergency Department (ED) | Cincinnati Children's Hospital Medical Center (CCHMC) Base ED | CCHMC Satellite ED | Children's National Medical Center (CNMC) Base ED | CNMC Satellite ED | The Children's Hospital Colorado Base ED | The Children's Hospital Colorado Satellite ED
Number analyzed (Participants) | 421622 | 409967 | 196300 | 376517 | 157802 | 316477 | 140776
number of visits | 421622 | 409967 | 196300 | 376517 | 157802 | 316477 | 140776

ADVERSE EVENTS:
Time Frame: January 2012- June 2016
Description: The study is without direct patient contact and utilizes only existing electronic health record data. The primary potential risk to subjects is improper disclosure of medical information.
Arm/Group | ED Patients
All-Cause Mortality (participants affected / at risk) | 0/2019461
Serious Adverse Events (participants affected / at risk) | 0/2019461
Other Adverse Events (participants affected / at risk) | 0/2019461

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-09-09): https://cdn.clinicaltrials.gov/large-docs/44/NCT01657344/Prot_SAP_000.pdf